CLINICAL TRIAL: NCT01464190
Title: An Open-label, Randomised, Active-controlled, Parallel Group, Multicentre Phase 3 Study to Investigate the Long-term Safety, Tolerability and Efficacy of PA21 Compared With Sevelamer Carbonate in Dialysis Patients With Hyperphosphataemia. Extension Study for Protocol PA-CL-05A (NCT01324128)
Brief Title: A Phase 3 Extension Study to Investigate the Long-term Safety, Tolerability and Efficacy of PA21, a Phosphate Binder in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA-CL-05B
Record Dates: First submitted 2011-09-12; First posted 2011-11-03 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: PA21; Phosphate Binder
MeSH Terms: interventions — Iron; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PA21 (Experimental)
  Interventions: Drug: PA21 (2.5 g tablet containing 500 mg iron)
- Sevelamer carbonate (Active Comparator)
  Interventions: Drug: Sevelamer carbonate

INTERVENTIONS:
Drug: PA21 (2.5 g tablet containing 500 mg iron) — Dose range of 5.0 g/day (2 tablets/day) to 15.0 g/day (6 tablets/day).
  Arms: PA21
Drug: Sevelamer carbonate — Film coated, compressed tablets. Dose range of 2.4 g/day (3 tablets/day) to 14.4 g/day (18 tablets/day).
  Arms: Sevelamer carbonate

SUMMARY:
This is a Phase 3, randomised, active controlled, multicentre extension study to investigate the long-term safety and efficacy of PA21, a phosphate binder, for control of hyperphosphataemia in dialysis patients. This is an extension study to PA-CL-05A (NCT01324128), subjects have already been enrolled and have been treated with study medication for at least 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed treatment in Protocol PA-CL-05A
* Written Informed Consent

Exclusion Criteria:

* Hyper/hypo calcemia; hyper intact parathyroid hormone (iPTH)
* Other significant medical conditions
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Floege, MD, Principal Investigator — Medizinische Klinik II
Locations (15):
- San Antonio, Texas, United States
- Medizinische Abteilung Nephrologie und Dialyse, Sankt Pölten, Austria
- CHU Sart Tilman, Liège, Belgium
- Clinical Hospital Center Rijeka, Rijeka, Croatia
- Hospital with Polyclinic Novy Jicin, Nový Jičín, Czechia
- KfH Nierenzentrum Berlin-Neukoelln, Berlin, Germany
- Vidzemes Hospital, Valmiera, Latvia
- JSC "Diaverum Clinics", Klaipėda, Lithuania
- Teaching Hospital no.1 of Medical University of Lodz, Lodz, Poland
- Dialmed Clinic SRL, Sibiu, Romania
- Kemerovo Regional hospital, Kemerovo, Russia
- Zvezdara Clinical Medical Center, Belgrade, Serbia
- St Augustines Hospital, Durban, South Africa
- Mykolayiv Regional Hospital, Mykolayiv, Ukraine
- Dorset County Hospital NHS Foundation Trust, Dorset, United Kingdom

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Sprague SM, Ketteler M, Covic AC, Floege J, Rakov V, Walpen S, Rastogi A. Long-term efficacy and safety of sucroferric oxyhydroxide in African American dialysis patients. Hemodial Int. 2018 Oct;22(4):480-491. doi: 10.1111/hdi.12663. Epub 2018 Apr 15. PMID 29656600

RESULTS

PARTICIPANT FLOW:
Groups:
- PA21: PA21 (2.5 g tablet). Dose range of 5.0 g/day (2 tablets/day) to 15.0 g/day (6 tablets/day)
- Sevelamer Carbonate: Sevelamer carbonate. Dose range of 2.4 g/day (3 tablets/day) to 14.4 g/day (18 tablets/day).
Period: Overall Study
Arm/Group | PA21 | Sevelamer Carbonate
Started | 391 | 268
Completed | 322 | 227
Not Completed | 69 | 41

BASELINE CHARACTERISTICS:
Population: For baseline characteristics, data from All Randomised patients was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | PA21 | Sevelamer Carbonate | Total
Number analyzed (Participants) | 391 | 268 | 659
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (13.20) | 55.6 (14.58) | 55.4 (13.77)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 296 | 190 | 486
  >=65 years | 95 | 78 | 173
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 102 | 273
  Male | 220 | 166 | 386
Region of Enrollment [Number; unit: participants]
  United States | 154 | 133 | 287
  Europe | 85 | 49 | 134
  Croatia | 16 | 8 | 24
  Russian Federation | 65 | 44 | 109
  Serbia | 37 | 18 | 55
  Ukraine | 32 | 15 | 47
  South Africa | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline and Levels at Each Time Point for Serum Phosphorus
Description: Endpoint is Week 28 or the latest available measurement after baseline when Week 28 data is missing.
Time Frame: Every 4 weeks from baseline to Week 28
Population: For the Primary Outcome, data from the Full Analysis Set for PA-CL-05B (FAS5B) was used. The FAS5B consists of all subjects who enrolled in PA-CL-05B, received at least 1 dose of PA-CL-05B medication, and had at least 1 efficacy assessment after the PA-CL-05B study entry visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA21 | Sevelamer Carbonate
Number analyzed (Participants) | 384 | 260
mg/dL
  Change from Baseline to Week 4 (n = 346, 236) | -0.2 (1.33) | -0.1 (1.47)
  Change from Baseline to Week 8 (n = 325, 238) | -0.2 (1.38) | 0.1 (1.56)
  Change from Baseline to Week 12 (n = 322, 242) | -0.0 (1.43) | 0.2 (1.55)
  Change from Baseline to Week 16 (n = 313, 228) | 0.0 (1.57) | 0.2 (1.75)
  Change from Baseline to Week 20 (n = 300, 221) | -0.0 (1.46) | 0.1 (1.44)
  Change from Baseline to Week 24 (n = 286, 208) | 0.1 (1.53) | 0.2 (1.78)
  Chnage from Baseline to Week 28 (n = 287, 210) | 0.2 (1.52) | 0.2 (1.76)
  Change from Baseline to Endpoint (n = 384, 260) | 0.1 (1.62) | 0.3 (1.79)

2. Primary Outcome: Change From Baseline and Levels at Each Time Point for Serum Calcium
Description: Endpoint is Week 28 or the latest available measurement after baseline when Week 28 data is missing.
Time Frame: Every 4 weeks from baseline to Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA21 | Sevelamer Carbonate
Number analyzed (Participants) | 384 | 260
mg/dL
  Change from Baseline to Week 4 (n = 346, 236 | -1.2 (12.07) | -0.8 (13.37)
  Change from Baseline to Week 8 (n = 325, 238) | -1.2 (12.30) | 1.5 (14.40)
  Change from Baseline to Week 12 (n = 321, 242) | 0.1 (12.94) | 1.9 (13.79)
  Change from Baseline to Week 16 (n = 313, 228) | 0.5 (14.04) | 2.0 (16.05)
  Change from Baseline to Week 20 (n = 300, 221) | 0.4 (13.24) | 1.6 (13.29)
  Change from Baseline to Week 24 (n = 284, 207) | 1.1 (13.57) | 2.2 (15.74)
  Change from Baseline to Week 28 (n = 286, 210) | 2.3 (13.52) | 2.3 (16.39)
  Change from Baseline to Endpoint (n = 365, 258) | 1.5 (13.86) | 2.9 (16.68)

3. Primary Outcome: Change From Baseline and Levels at Each Time Point for Serum Intact Parathyroid Hormone (iPTH)
Description: Endpoint is Week 28 or the latest available measurement after baseline when Week 28 data is missing.
Time Frame: Every 4 weeks from baseline to Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PA21 | Sevelamer Carbonate
Number analyzed (Participants) | 384 | 260
pg/mL
  Change from Baseline to Week 4 (n = 365, 252) | 11.8 (177.39) | 25.9 (186.42)
  Change from Baseline to Week 8 (n = 362, 258) | 8.6 (204.39) | 40.8 (201.18)
  Change from Baseline to Week 12 (n = 352, 252) | 28.9 (315.81) | 64.1 (204.11)
  Change from Baseline to Week 16 (n = 341, 241) | 54.5 (352.92) | 52.3 (210.35)
  Change from Baseline to Week 20 (n = 334, 236) | 28.0 (233.13) | 72.1 (228.03)
  Change from Baseline to Week 24 (n = 320, 226) | 27.7 (271.31) | 79.6 (253.65)
  Change from Baseline to Week 28 (n = 310, 222) | 53.0 (287.19) | 71.5 (278.03)
  Change from Baseline to Endpoint (n = 381, 260) | 52.3 (273.14) | 67.5 (270.06)

ADVERSE EVENTS:
Description: For the serious adverse event (SAE) and adverse event (AE) listings, data from the Safety Set for PA-CL-05B (SS5B). The SS5B consists of all enrolled subjects who had taken at least 1 dose of PA-CL-05B study medication.
Arm/Group | PA21 | Sevelamer Carbonate
Serious Adverse Events (participants affected / at risk) | 78/391 | 52/267
Other Adverse Events (participants affected / at risk) | 208/391 | 169/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA21 (N=391) | Sevelamer Carbonate (N=267)
Abdominal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Aneurysm ruptured (Vascular disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Arteriovenous graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (4) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (4) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Device occlusion (General disorders) | 1 (1) | 0 (0)
Diabetic foot (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 4 (5) | 6 (6)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 2 (2) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 4 (4) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypocoagulable state (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 6 (6)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Renal cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cyst ruptured (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 2 (2)
Shunt malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Infections and infestations) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA21 (N=391) | Sevelamer Carbonate (N=267)
Anaemia (Blood and lymphatic system disorders) | 15 (16) | 15 (17)
Diarrhoea (Gastrointestinal disorders) | 32 (43) | 15 (19)
Headache (Nervous system disorders) | 20 (28) | 8 (19)
Hyperkalaemia (Metabolism and nutrition disorders) | 17 (31) | 16 (28)
Hyperparathyroidism secondary (Endocrine disorders) | 15 (15) | 23 (25)
Hyperphosphataemia (Metabolism and nutrition disorders) | 47 (73) | 29 (47)
Hypertension (Vascular disorders) | 38 (53) | 20 (29)
Hypophosphataemia (Metabolism and nutrition disorders) | 22 (26) | 14 (14)
Hypotension (Vascular disorders) | 19 (37) | 21 (38)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26 (39) | 16 (20)
Nausea (Gastrointestinal disorders) | 23 (26) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may not present or publish partial or complete study results individually. Any manuscript or abstract proposed by the Investigators must be reviewed and approved in writing by Vifor Pharma before submission for publication. Names of all Investigators participating in the study will be included in the publication.